CLINICAL TRIAL: NCT04841161
Title: Development of an Intelligent Balance Training System Providing Weight-bearing Feedback Via Force Platform to Improve Sit-to-stand, Dynamic Weight-shifting and Standing Performance in Stroke Patients
Brief Title: Development of an Intelligent Balance Training System Providing Weight-bearing Feedback in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-F(II)-20150033
Record Dates: First submitted 2021-03-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Other): The healthy adults who have not any neurological, musculoskeletal or rhematogical disease, a history of orthopedic surgery on spine or lower extremity. Their age should be ranged between 20 - 75 years.
  Interventions: Behavioral: Balance function, gait ability, weight- distribution and weight-shifting
- Stroke subjects (Experimental): Stroke patients were included if they were: (1) diagnosed with unilateral ischemic or hemorrhagic stroke; (2) a minimum of six months post stroke ; (2) able to stand without support for 1 minutes; (3) able to understand and follow verbal instructions. and (4) medically stable with physician release.
  Interventions: Behavioral: Balance function, gait ability, weight- distribution and weight-shifting; Behavioral: Weight- distribution and weight-shifting training program

INTERVENTIONS:
Behavioral: Balance function, gait ability, weight- distribution and weight-shifting — Healthy adults and stroke patients accepted two measurements within a week. Balance function, gait ability, weight- distribution and weight-shifting during sit-to-stand, quite standing, and weight-shifting toward the forward foot.
Behavioral: Weight- distribution and weight-shifting training program — The stroke patients received a weight-shifting training program , 30 minutes/time, 2-5 days a week for 2-3 weeks(8 sessions). After training, they accepted a post-test within a week.
  Arms: Stroke subjects

SUMMARY:
The sit-to-stand and dynamic weight-shifting ability of stroke patients is highly associated with walking performance. Therefore, in order to improve the dynamic weight-shifting ability in sit-to-stand and parallel or tandem standing, a real-time visual or auditory feedback is used in our design to allow patients to realize the weight-bearing condition (by using load cells) in both sound and affected legs immediately. It can help patients to learn to control muscle to shift weight effectively which will improve patients' walking performance. By integrating physical therapy planning with electro-mechanical technology, the goal of this study is to develop a standing balance training system by requiring patients to control their center of pressure (COP) in performing sit-to-stand and maintain a standing posture via the use of their core and lower extremity musculature.

DETAILED DESCRIPTION:
1. Written informed consent must be obtained before any study specific procedures are undertaken.

1. For healthy group: Participants will be recruited from the staffs and students in Kaohsiung Medical University (including Learning University), and healthy families of CVA patients in the university affiliated hospital.
2. For stroke (CVA) group: We will ask the physical therapists in the university affiliated hospital to nominate the potential CVA participants . The physicians will determine if they would meet the inclusion criteria before participating the present study.

2. The process of the experiment (brief describe)

1. Written informed consent must be obtained before any study specific procedures are undertaken.
2. Subjects who are recruited to participate in this experiment should provide the personal information forms first (ex: sex, age, height, weight, post-stroke duration, stroke type, hemiplegic side, ambulation devices etc.). Then, assessment (PASS, Berg Balance Scale, Timed Up and Go) will be conducted by a physical therapist at baseline.
3. While the stroke patients after completing the 4 -times, and 8-times training program, the above-mentioned assessment conducted again by the same physical therapist. The healthy will not receive balance training, thus .only receive one assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults

   a. Their age should be ranged between 20 - 75 years
2. Stroke patients

   1. diagnosed with unilateral ischemic or hemorrhagic stroke
   2. a minimum of six months post stroke
   3. able to stand without support for 1 minutes
   4. medically stable with physician release

Exclusion Criteria:

1. Healthy adults

   1. neurological diseases
   2. musculoskeletal diseases
   3. rheumatic diseases
   4. history of orthopedic surgery on spine or lower extremity
2. Stroke patients

   1. other injuries or illnesses that affect standing or walking

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Changes in performance of weight distribution after 8 sessions intervention | The assessments will be conducted before and after intervention (4 Weeks, 8 Sessions)
  By using the force plate to record the ground reaction force and then to obtain weight distribution while performing the sit to stand activity
Changes in performance of standing balance after 8 sessions intervention | The assessments will be conducted before and after intervention (4 Weeks, 8 Sessions)
  By using the force plate to obtain displacements of the center of pressure (COP) while standing and weight transfer
Changes in performance of static and dynamic balance after 8 sessions intervention | The assessments will be conducted before and after intervention (4 Weeks, 8 Sessions)
  By using the Postural Assessment Scale of Stroke (PASS) to assess and monitor postural control. The PASS consists of 2 sections with a 4-point scale to describe each task. The total score ranges from 0 - 36.
Changes in performance of balance function after 8 sessions intervention | The assessments will be conducted before and after intervention (4 Weeks, 8 Sessions)
  By using the Berg Balance Scale to assess balance function. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4during a series of predetermined tasks. The total score ranges from 0 - 56.
Changes in performance of dynamic balance after 8 sessions intervention | The assessments will be conducted before and after intervention (4 Weeks, 8 Sessions)
  By using Timed Up and Go Test (TUG) to assess fall risk and measure the progress of balance. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jiun Liaw, Study Director — Kaohsiung Medical University Department of Physical Therapy Associate Professor
Locations (1):
- Li-Jiun Liaw, Kaohsiung City, Sanmin Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No
Currently in the submission stage ,and then share with other researchers after publication